CLINICAL TRIAL: NCT03013309
Title: An Individually Tailored, Family-Centered Intervention for Childhood Obesity: Connecting Services in Pediatric Primary Healthcare, the Home and the Community
Brief Title: Raising Healthy Children: A Hybrid Trial of the Family Check-Up 4 Health in Primary Care
Acronym: FCU4Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Northwestern University (Other); University of Washington (Other); University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1U18DP006255-01 (NIH)
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Clinical Trial
Keywords: Hybrid; Implementation; Effectiveness; Parent training; Fidelity; Cost-Effectiveness; Primary Care
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Receives the Family Check-Up 4 Health
  Interventions: Behavioral: Family Check-Up 4 Health
- Control (Experimental): Receives Treatment as Usual
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Family Check-Up 4 Health — A parent-training intervention to improve child health and prevent/manage obesity
  Other Names: FCU4Health
  Arms: Intervention
Other: Treatment as usual — Treatment as usual
  Arms: Control

SUMMARY:
This study is a hybrid implementation-effectiveness trial of the Family Check-Up 4 Health (FCU4Health), an adapted version of the Family Check-Up, in pediatric primary care. Patients will be recruited based on their BMI as documented in the Electronic Health Record (EHR) and randomized to receive the FCU4Health or Treatment as Usual.

DETAILED DESCRIPTION:
The FCU4Health is an assessment-driven, Motivational Interviewing (MI) based, parent training program. Parents and children complete a comprehensive assessment, including questionnaire and observation data. The FCU4Health coordinator reviews the assessment results with the parents, using MI strategies to create a tailored plan to address family needs. This plan may include referrals to community resources or parenting modules that focus on family management.

ELIGIBILITY:
Inclusion Criteria:

* BMI at or above 85% tile for age and gender

Exclusion Criteria:

-

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
BMI | The investigators will examine trajectories based on 4 assessments over one year
  BMI

SECONDARY OUTCOMES:
Body Composition | The investigators will examine trajectories based on 4 assessments over one year
  % Body fat
EuroQol-5D-5Level-Youth (EQ-5D-5L-Y) | The investigators will examine trajectories based on 4 assessments over one year
  Quality of life
PedsQL | The investigators will examine trajectories based on 4 assessments over one year
  Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Cady Berkel, Ph.D., Principal Investigator — Arizona State University
Locations (3):
- United States (3):
  - Terros Health, Phoenix, Arizona
  - Valle del Sol, Phoenix, Arizona
  - Phoenix Children's Hospital, Phoenix, Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berkel C, Knox DC, Flemotomos N, Martinez VR, Atkins DC, Narayanan SS, Rodriguez LA, Gallo CG, Smith JD. A machine learning approach to improve implementation monitoring of family-based preventive interventions in primary care. Implement Res Pract. 2023 Jul 25;4:26334895231187906. doi: 10.1177/26334895231187906. eCollection 2023 Jan-Dec. PMID 37790171
- [Derived] Harris A, Jordan N, Carroll AJ, Graham AK, Wilson C, Wilson FA, Berkel C, Smith JD. A budget impact analysis of cost to implement a whole child health focused, family-based intervention in primary care for children with elevated BMI. Implement Sci Commun. 2023 Jun 5;4(1):59. doi: 10.1186/s43058-023-00429-z. PMID 37277878
- [Derived] Smith JD, Carroll AJ, Fu E, Berkel C. Baseline Targeted Moderation in a Trial of the Family Check-Up 4 Health: Potential Explanations for Finding Few Practical Effects. Prev Sci. 2023 Feb;24(2):226-236. doi: 10.1007/s11121-021-01266-z. Epub 2021 Jun 22. PMID 34159507
- [Derived] Berkel C, Fu E, Carroll AJ, Wilson C, Tovar-Huffman A, Mauricio A, Rudo-Stern J, Grimm KJ, Dishion TJ, Smith JD. Effects of the Family Check-Up 4 Health on Parenting and Child Behavioral Health: A Randomized Clinical Trial in Primary Care. Prev Sci. 2021 May;22(4):464-474. doi: 10.1007/s11121-021-01213-y. Epub 2021 Mar 14. PMID 33715136
- [Derived] Smith JD, Berkel C, Jordan N, Atkins DC, Narayanan SS, Gallo C, Grimm KJ, Dishion TJ, Mauricio AM, Rudo-Stern J, Meachum MK, Winslow E, Bruening MM. An individually tailored family-centered intervention for pediatric obesity in primary care: study protocol of a randomized type II hybrid effectiveness-implementation trial (Raising Healthy Children study). Implement Sci. 2018 Jan 15;13(1):11. doi: 10.1186/s13012-017-0697-2. PMID 29334983